CLINICAL TRIAL: NCT00775372
Title: An Open Label, Balanced, Randomised, Two-Treatment, Four-Period, Two- Sequence, Single-Dose, Crossover Fully Replicated, Bioavailability Study on Clarithromycin Formulations Comparing Clarithromycin 250 mg/5 mL Powder for Oral Suspension of Ranbaxy Laboratories With Biaxin® Granules 250 mg/5 mL Oral Suspension in Healthy, Adult,Human, Male Subjects Under Fed Conditions.
Brief Title: Bioequivaelnce Study of Clarithromycin 250 mg/5 mL Powder for Oral Suspension Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CPU-N-015/CLARI-250/05
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence study of clarithromycin 250mg/5mL powdder
MeSH Terms: interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): clarithromycin 250 mg/5 mL powder for oral suspension of Ranbaxy Laboratories
  Interventions: Drug: Clarithromycin 250mg/5mL
- 2 (Active Comparator): Biaxin® granules 250 mg/5 mL oral suspension
  Interventions: Drug: Clarithromycin 250mg/5mL

INTERVENTIONS:
Drug: Clarithromycin 250mg/5mL

SUMMARY:
To compare the single-dose oral bioavailability of clarithromycin 250 mg/5 mL powder for oral suspension of Ranbaxy Laboratories with Biaxin 250 mg/5 mL granules for oral suspension in healthy, adult, human, male subjects under fed conditions

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomised, two-treatment, four-period, two-sequence, single-dose, crossover fully replicated, bioavailability study on clarithromycin formulations comparing clarithromycin 250 mg/5 mL powder for oral suspension of Ranbaxy Laboratories with Biaxin® granules 250 mg/5 mL oral suspension in healthy, adult, human, male subjects under fed conditions

A single oral dose of clarithromycin 250 mg/5 mL was administered during each period under supervision of a trained Medical Officer.

During the course of study, the safety parameters including vital signs, physical examination, medical history, clinical laboratory and safety tests (haematology, biochemical parameters) were assessed and, clinical laboratory safety tests (hematology & biochemical parameters) were performed again at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Be in the age range of 18-45 years.
* Be neither overweight nor underweight for his/her height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
* Have voluntarily given written informed consent to participate in this study.
* Be of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.

Exclusion Criteria:

* History of allergy to clarithromycin, erythromycin and related macrolides.
* History of severe diarrhoea within 2 weeks preceding Day 1 of this study.
* Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations
* Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
* Presence of values which are significantly different from normal reference ranges (as defined in Appendix 5) and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.
* Positive for urinary screen testing of drugs of abuse (opiates or cannabinoids)
* Presence of values which are significantly different from normal reference ranges (as defined in Appendix 5) and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
* Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), glucose (positive) or protein (positive).
* Clinically abnormal ECG or Chest X-ray.
* QTc interval beyond normal limits
* History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes or glaucoma.
* History of any psychiatric illness which may impair the ability to provide written informed consent.
* Regular smokers who smoke more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
* History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or have difficulty in abstaining for the duration of each study period.
* Use of any enzyme modifying drugs within 30 days prior to Day 1 of this study.
* Participation in any clinical trial within 12 weeks preceding Day 1 of this study.
* A haemoglobin concentration of less than 7 % of lower limit of reference range e.g. 13 gm % for reference range of 14-18 gm at screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2005-09; Primary Completion 2005-10 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Ranbaxy Research Laboratories, Gurgaon, Haryana, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html